CLINICAL TRIAL: NCT04475874
Title: Efficacy of Active Stretching Exercises on Symptoms of Primary Dysmenorrhea
Brief Title: Stretching Exercises on Symptoms of Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, ZIZI MOHAMMED IBRAHIM ALI, ASSOCIATE PROF, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPTPNU
Record Dates: First submitted 2020-07-12; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- supervised stretching exercises :group A (Active Comparator): The intervention group A practiced a 30 to 45-minute supervised active stretching program three times a week for four weeks
  Interventions: Other: supervised stretching exercises
- non-supervised active stretching home program: group B (Active Comparator): practiced non-supervised active stretching home program
  Interventions: Other: non-supervised active stretching home program
- Standard of care: group c (No Intervention): control group

INTERVENTIONS:
Other: supervised stretching exercises — 30 to 45-minute supervised active stretching program by a trained physical therapist, three times a week for four weeks starting with a warmup of 5 minutes on a stationary bicycle, half jumping jacks and torso rotations
  Other Names: home program stretching exercises
  Arms: supervised stretching exercises :group A
Other: non-supervised active stretching home program — non supervised 30 to 45-minute supervised active stretching program three times a week for four weeks starting with a warmup of 5 minutes on a stationary bicycle, half jumping jacks and torso rotations
  Other Names: home program of stretching exercises
  Arms: non-supervised active stretching home program: group B

SUMMARY:
The purpose of this study was to assess the effect of active stretching exercises on reducing pain and the quality of life during menstrual cycle in young adult females.

DETAILED DESCRIPTION:
Thirty females with primary dysmenorrhea, aging between 18 to 23 years with BMI of 20-29.9 kg/m2, have a regular menstrual cycle length 28-30 day and cycle bleed from 3 to 7 days, were randomly assigned into three equal groups; two interventions groups (supervised and non-supervised active stretching exercise program) and one control group. The intervention group A practiced a 30 to 45-minute supervised active stretching program three times a week for four weeks, while the other intervention group B practiced non-supervised active stretching home program and the control group C . Visual Analog Scale (VAS) was used to measure pain intensity, and Verbal Multidimensional System (VMS) for measuring menstruation characteristics and the effect of pain on quality of life, before (pre) as well as after (post) 4 weeks at the end of the study .

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20-29.9 kg/m2,
* regular menstrual cycle
* length 28-30 day
* cycle bleed from 3 to 7 days,

Exclusion Criteria:

* contraindication to stretching exercise
* taking any hormonal medications:
* smoker

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline at pain intensity 4 weeks after
  Visual Analog Scale measures pain intensity it is a unidimensional measure of pain intensity The classification of VAS was done according to pain scores (mild: 1-3 Moderate: 4-7 Severe: 8-10)

SECONDARY OUTCOMES:
Verbal Multidimensional System(VMS) | Change from Baseline amenstruation characteristics 4 weeks after
  Verbal Multidimensional System which is a grading system from zero to three and used to evaluate menstruation characteristics including the working ability, the systemic symptoms and analgesia requirement in order to decrease pain with dysmenorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Zizi Mohammed Ibrahim Ali, Riyadh, Nnjkjk, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No